CLINICAL TRIAL: NCT05979636
Title: Effect of Toothpaste Containing Novamin on Streptococcous Mutans Count in Dental Plaque of High Caries Risk Children (Randomized Controlled Clinical Trial)
Brief Title: Novamin on Streptococcus Mutans Count in Dental Plaque of High Caries Risk Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0286-09/2021
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Dental Plaque; Dental Caries
MeSH Terms: conditions — Dental Plaque; Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Novamin containing toothpaste
- Control group (Active Comparator)
  Interventions: Other: Fluoride containing toothpaste

INTERVENTIONS:
Other: Novamin containing toothpaste — children's teeth will be brushed using Novamin containing toothpaste.
  Arms: Test group
Other: Fluoride containing toothpaste — children's teeth will be brushed using Fluoride containing toothpaste.
  Arms: Control group

SUMMARY:
Inhibition of streptococcus mutans can be effective to prevent caries in high caries-risk children. The aim of the study is to evaluate the effect of Novamin on streptococcus mutans in the plaque of high caries-risk children.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy children.
* No erupting first permanent molars.
* High caries risk children; Have visible cavities or have a visible plaque on their teeth.
* Cooperative (Positive or definitely positive), according to Frankl's Behavior Rating Scale

Exclusion Criteria:

* History of intake of antibiotics for the past 3-4 weeks.
* History of professional fluoride treatment over 2 weeks before the study.
* Children with tooth structure defects.
* Children unable to return for recall visits

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in bacterial count in dental plaque | 1 week, 2 weeks and 4 weeks
  The samples will be collected from all children in the study and the level of S.mutans will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt